CLINICAL TRIAL: NCT03876977
Title: Robotic Decompression of the Pudendal Nerve in Pudendal Neuralgia: A Randomized Controlled Trial
Brief Title: Robotic Decompression of the Pudendal Nerve in Pudendal Neuralgia
Acronym: ERIS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitments difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7253
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Robotic Decompression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive (No Intervention): Neuropathic drugs Pudendal infiltration
- Robotic laparoscopic decompression (Experimental): Robotic laparoscopic decompression of pudendal nerve entrapment.
  Interventions: Procedure: Robotic laparoscopic decompression of pudendal nerve entrapment

INTERVENTIONS:
Procedure: Robotic laparoscopic decompression of pudendal nerve entrapment — Robotic laparoscopic decompression of pudendal nerve entrapment.
  Transperitoneal Laparoscopic Robotic assistance
  Arms: Robotic laparoscopic decompression

SUMMARY:
Primary purpose:

Show the pain improvement 3-month after robotic laparoscopic pudendal nerve decompression for pudendal neuralgia.

Primary outcomes:

Pain evaluated on a VAS before surgery and 3-month after surgery or surveillance Improvement is considered if pain decreased by at least 3/10 points on the VAS.

Secondary purposes:

* improvement of quality of life
* study of MRI performance to predict pudendal nerve entrapment topography
* show the feasibility and safety of robotic pudendal nerve decompression

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70 years old
* Pudendal neuralgia according to Nantes criteria
* pudendal nerve entrapment reachable with robotic transperitoneal approach

Exclusion Criteria:

* bilateral pain
* history of pain ≥ 18 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-08-08 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Collection of the maximum pain intensity on a numerical scale (EN), calculated on 10 points. (0 no pain -10 extreme pain ) | 3-months after surgery or surveillance
  Collection of the maximum pain intensity on a numerical scale (EN), calculated on 10 points.
  Daily collection by the patient over 1 week in real life conditions. Achievement of an average of the scores over 1 week.

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'urologie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No